CLINICAL TRIAL: NCT07390747
Title: A Phase 1, Randomized, Double-blind, Placebo-Controlled Study to Evaluate the Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of a Single Subcutaneous Administration of SHR-2173 in Healthy Participants
Brief Title: A Trial of SHR-2173 in Healthy Volunteers
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Atridia Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-2173-106
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Immunology

STUDY DESIGN:
Intervention Model Description: Single dose of SHR-2173 will be administered subcutaneously
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-2173 single dose (Experimental): Single dose of SHR-2173 given subcutaneously
  Interventions: Drug: SHR-2173 Injection/SHR-2173 placebo
- SHR-2173 placebo single dose (Experimental): Single dose of SHR-2173 placebo given subcutaneously
  Interventions: Drug: SHR-2173 Injection/SHR-2173 placebo

INTERVENTIONS:
Drug: SHR-2173 Injection/SHR-2173 placebo — Single dose SHR-2173 injection or matching placebo given subcutaneously

SUMMARY:
The purpose of this study is to assess safety, PK, Pharmacodynamic and immunogenicity profile of a single dose of SHR-2173 in healthy participants

ELIGIBILITY:
Main inclusion criteria

1. Healthy white participants.
2. Ability to understand the trial procedures and possible adverse events, volunteer to participate in the trial, and provide written informed consent, be able to comply with all the requirements, and able to complete the study.
3. Male aged between 18 to 45 years of age (inclusive)
4. Women with body weight ≥ 45.0 kg, men with body weight ≥ 50.0 kg, body mass index (BMI) between 19.0 and 30.0 kg/m2 (inclusive) at screening.
5. Men and WOCBP must agree to take highly effective contraceptive methods

Main exclusion Criteria

1. History or evidence of clinically significant disorders.
2. Individuals with a history of drug allergies, specific allergies, or known history or suspected of being allergic to the study or same class drug or any component of it.
3. Receipt of medical devices or another investigational drug within 3 months or 5 half-lives, whichever is longer prior to screening.
4. The injection site has abnormalities or is deemed by the investigator as unsuitable for subcutaneous injection.
5. History of excessive smoking in the past 1 month prior to screening
6. History of illicit or prescription drug abuse or addiction within 1 year of screening, or positive urine drug screen at baseline.
7. Any other circumstances (e.g., not suitable for venous access) or laboratory abnormality that, in the investigator's judgment, may increase the risk to the participant, or be associated with the participant's participation in and completion of the study or could preclude the evaluation of the participant's response.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics - Cmax | Day 71
  Maximum observed plasma concentration (Cmax)
Pharmacokinetics - AUC₀-t | Day 71
  Area under the plasma concentration-time curve from time 0 to the last measurable concentration (AUC₀-t)
Pharmacokinetics - AUC₀-inf | Day 71
  Area under the plasma concentration-time curve from time 0 extrapolated to infinity (AUC₀-inf)
Pharmacokinetics - Tmax | Day 71
  Time to reach maximum observed plasma concentration (Tmax)
Pharmacokinetics - t½ | Day 71
  Terminal elimination half-life (t½)
Immunogenicity - Anti-Drug Antibody (ADA) | Day 71
  Incidence and onset time of anti-drug antibody (ADA)

SECONDARY OUTCOMES:
Safety and Tolerability Based on Incidence and Severity of Treatment Emergent Adverse Events | Day 71
  Number of participants with Adverse events and Serious adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Veritus Research, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Undecided